CLINICAL TRIAL: NCT04707976
Title: A Randomized Controlled Trial Comparing the Efficacy of Transanal Irrigation With Navina Smart Versus Standard Bowel Care in Patients With Multiple Sclerosis
Brief Title: Comparing Transanal Irrigation With Navina Smart vs. Standard Bowel Care in Patients With Multiple Sclerosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wellspect HealthCare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NAV-0006
Record Dates: First submitted 2020-10-22; First posted 2021-01-13 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Neurogenic Bowel (Disorder); Fecal Constipation; Fecal Incontinence; Multiple Sclerosis
MeSH Terms: conditions — Neurogenic Bowel; Fecal Incontinence; Multiple Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Navina Smart (Experimental): An electronic medical device to perform transanal irrigation. Treatment period 8 weeks.
  Interventions: Device: Navina Smart
- Standard Bowel Care (Active Comparator): Supportive bowel care without using irrigation.
  Interventions: Other: Standard Bowel Care

INTERVENTIONS:
Device: Navina Smart — CE-marked NavinaTM Smart including Navina Smart App.
  Arms: Navina Smart
Other: Standard Bowel Care — Bowel care will be scheduled at least every 2nd day according to a defined study specific standard bowel care protocol. Diet, fluids, abdominal massage, regular physical activity and medications will be used if non-interventional treatment is insufficient.
  Arms: Standard Bowel Care

SUMMARY:
A randomized, superiority, controlled, interventional, prospective, multicentre, post-market study of TAI with Navina™ Smart versus Standard Bowel Care performed in a population of 92 subjects suffering from Multiple Sclerosis and confirmed Neurogenic Bowel Dysfunction. The study is expected to last for a total of 8 weeks per subject with two scheduled site visits.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, subjects must fulfil all of the following criteria:

1. Provision of informed consent.
2. Female or male aged 18 years or above.
3. Established diagnosis of MS according to McDonald criteria.
4. Patients with bowel symptoms post-dating and related to a diagnosis of MS.
5. Patients suffering from NBD symptoms defined by Wexner feacal incontinence score ≥10 and/or Cleveland Clinic constipation score ≥10 confirmed at Baseline.
6. Only TAI treatment naïve patient (not having previously used any particular TAI system).
7. Judged eligible for TAI as per standardized treatment pathway.
8. Able to read, write and understand information given to them regarding the study.

Exclusion Criteria:

Any of the following is regarded as a criterion for exclusion from the study:

1. Any confirmed or suspected diagnosis of anal or colorectal stenosis, active inflammatory bowel disease, acute diverticulitis, severe diverticulosis, colorectal cancer, ischemic colitis, history of life-threatening autonomic dysreflexia, bleeding disorders, unspecified peri-anal conditions.
2. Untreated rectal impaction.
3. Other significant neurological diseases (defined as all neurological diseases except for minor functional neurological syndromes or non-MS related neuro complications).
4. Opioid consumption ≤24 hours prior enrolment.
5. Previous colorectal surgery (including haemorrhoidectomy and fistulotomy), sphincter injury, perianal sepsis, rectal prolapse.
6. Performed endoscopic polypectomy within 4 weeks prior enrolment.
7. Ongoing, confirmed pregnancy or lactation.
8. Any neuromodulation that can affect the pelvic organ function.
9. Ongoing, symptomatic Urinary Tract Infection (UTI) at enrolment (defined as a positive urine culture of ≥10^3 CFU/ml of ≥1 bacterial species and presence of symptoms or signs compatible with UTI with no other identified source of infection).*
10. Current treatment with anticoagulants (exception acetylsalicylic acid or clopidogrel).
11. Current treatment with long-term systemic steroid medication (exception inhalation agents and/or local topical treatment).
12. Current treatment of prokinetics.
13. Involvement in the planning and conduct of the study (applies to both Wellspect HealthCare and site personnel).
14. Previous enrolment in the present study.
15. Simultaneous participation in another clinical study that may interfere with the present study as judged by the investigator.
16. Expected severe non-compliance to protocol as judged by the investigator.
17. Any other condition, as judged by the investigator, which might make follow-up or investigations inappropriate.
18. Any patient that according to the Declaration of Helsinki is unsuitable for enrolment.
19. Agranulocytosis (<0.5 10^9 / L) [Only applicable for Switzerland].

    * If symptoms and signs compatible with UTI is present but no urine culture test has been performed yet, a test should be performed, and the result received prior evaluating if the subject is eligible for study participation. After successful and completed treatment of a UTI, the subject may be rescheduled for Visit 1 in order to re-evaluate study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Change in fecal incontinence score. | 8 weeks
  Relative change in Wexner fecal incontinence score at 8 weeks relative to Baseline in the TAI arm, compared to the SBC arm.
Change in fecal constipation score | 8 weeks.
  Relative change in Cleveland Clinic constipation score at 8 weeks relative to Baseline in the TAI arm, compared to the SBC arm.

SECONDARY OUTCOMES:
Efficacy of TAI with Navina Smart vs. SBC | 4 weeks
  Absolute change in Wexner fecal incontinence score at 4 weeks relative to Baseline in the TAI arm, compared to the SBC arm.
Efficacy of TAI with Navina Smart vs. SBC | 8 weeks
  Absolute change in Wexner fecal incontinence score at 8 weeks relative to Baseline in the TAI arm, compared to the SBC arm.
Efficacy of TAI with Navina Smart vs. SBC | 4 weeks
  Absolute change in Cleveland Clinic constipation score at 4 relative to Baseline in the TAI arm, compared to the SBC arm.
Efficacy of TAI with Navina Smart vs. SBC | 8 weeks
  Absolute change in Cleveland Clinic constipation score at 4 relative to Baseline in the TAI arm, compared to the SBC arm.
Efficacy of TAI with Navina Smart vs. SBC | 4 weeks
  Relative change in Wexner fecal incontinence score at 4 weeks relative to Baseline in the TAI arm, compared to the SBC arm.
Efficacy of TAI with Navina Smart vs. SBC | 8 weeks
  Relative change in Wexner fecal incontinence score at 4 weeks relative to Baseline in the TAI arm, compared to the SBC arm.
Efficacy of TAI with Navina Smart vs. SBC | 4 weeks
  Relative change in Cleveland Clinic constipation score at 4 weeks relative to Baseline in the TAI arm, compared to the SBC arm
Efficacy of TAI with Navina Smart vs. SBC | 8 weeks
  Relative change in Cleveland Clinic constipation score at 4 weeks relative to Baseline in the TAI arm, compared to the SBC arm
Change in perception of impact of bowel symptoms on QoL | 8 weeks
  Relative change of impact on bowel-related QoL between baseline and 8 weeks in the TAI arm, compared to the SBC arm, as measured by a single question.
Change in NBD symptoms | 4 weeks and 8 weeks
  Absolute and relative change in NBD score between Baseline and 4 and 8 weeks in the Navina arm, compared to the SBC arm.
Change in bladder specific QoL | 8 weeks
  Absolute and relative change in SF-Qualiveen questionnaire between Baseline and 8 weeks in the TAI arm, compared to the SBC arm.
Study therapy adherence | 4 weeks and 8 weeks
  Number of subjects using Navina Smart or SBC at 4 weeks and 8 weeks treatment, as measured by a single question.
Frequency of UTI | 8 weeks
  Number of UTIs requiring antibiotic treatment 8 weeks prior study start (Baseline) and at 8 weeks after treatment (Visit 2), as reported by subject.
Navina Smart: Correlation APP/irrigation parameters | Up to 3 weeks
  Volume correlation with Anorectal Physiology Parameters (APPs) up to 3 weeks from baseline in subjects who perform the anorectal physiology test, treated with Navina Smart, and using the Navina Smart App.
Navina Smart: Correlation APP/irrigation parameters | 4 weeks
  Volume correlation with Anorectal Physiology Parameters (APPs) after 4 weeks in subjects who perform the anorectal physiology test, treated with Navina Smart, and using the Navina Smart App
Navina Smart: Correlation APP/irrigation parameters | 8 weeks.
  Volume correlation with Anorectal Physiology Parameters (APPs) after 8 weeks in subjects who perform the anorectal physiology test, treated with Navina Smart, and using the Navina Smart App
Navina Smart: Correlation APP/irrigation parameters | Up to 3 weeks
  Frequency of irrigations correlation with Anorectal Physiology Parameters (APPs) up to 3 weeks from baseline in subjects who perform the anorectal physiology test, treated with Navina Smart, and using the Navina Smart App
Navina Smart: Correlation APP/irrigation parameters | 4 weeks
  Frequency of irrigations correlation with Anorectal Physiology Parameters (APPs) after 4 weeks in subjects who perform the anorectal physiology test, treated with Navina Smart, and using the Navina Smart App.
Navina Smart: Correlation APP/irrigation parameters | 8 weeks.
  Frequency of irrigations correlation with Anorectal Physiology Parameters (APPs) after 8 weeks in subjects who perform the anorectal physiology test, treated with Navina Smart, and using the Navina Smart App.
Navina Smart: Correlation APP/irrigation parameters | Up to 3 weeks
  Balloon inflation correlation with Anorectal Physiology Parameters (APPs) up to 3 weeks from baseline in subjects who perform the anorectal physiology test, treated with Navina Smart, and using the Navina Smart App
Navina Smart: Correlation APP/irrigation parameters | 4 weeks
  Balloon inflation correlation with Anorectal Physiology Parameters (APPs) after 4 weeks in subjects who perform the anorectal physiology test, treated with Navina Smart, and using the Navina Smart App
Navina Smart: Correlation APP/irrigation parameters | 8 weeks.
  Balloon inflation correlation with Anorectal Physiology Parameters (APPs) after 8 weeks in subjects who perform the anorectal physiology test, treated with Navina Smart, and using the Navina Smart App.
Navina Smart: Correlation anorectal APP/irrigation parameters between responders/non-responders | Up to 3 weeks
  Correlation between Anorectal Physiology Parameters (APPs), irrigations parameters (volume/frequency of irrigation and balloon inflation) and outcome of TAI treatment between responders versus non-responders in subjects who perform the anorectal physiology test, treated with Navina Smart, and using the Navina Smart App from baseline to 3 weeks. A responder is defined as an improvement equal to the 25th percentile of the change in Cleveland Clinic Constipation score when using TAI with Navina Smart.
Navina Smart: Correlation anorectal APP/irrigation parameters between responders/non-responders | 4 weeks
  Correlation between Anorectal Physiology Parameters (APPs), irrigations parameters (volume/frequency of irrigation and balloon inflation) and outcome of TAI treatment between responders versus non-responders in subjects who perform the anorectal physiology test, treated with Navina Smart, and using the Navina Smart App for 4 weeks. A responder is defined as an improvement equal to the 25th percentile of the change in Cleveland Clinic Constipation score when using TAI with Navina Smart.
Navina Smart: Correlation anorectal APP/irrigation parameters between responders/non-responders | 8 weeks
  Correlation between Anorectal Physiology Parameters (APPs), irrigations parameters(volume/frequency of irrigation and balloon inflation) and outcome of TAI treatment between responders versus non-responders in subjects who perform the anorectal physiology test, treated with Navina Smart, and using the Navina Smart App for 8 weeks. A responder is defined as an improvement equal to the 25th percentile of the change in Cleveland Clinic Constipation score when using TAI with Navina Smart.

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Schürch, Prof., Principal Investigator — Département des neurosciences cliniques Centre Hospitalier Universitaire Vaudois (CHUV); Lausanne; Bonaventura Casanova, Dr., Principal Investigator — Unidad de Esclerosis Multiple - Servicio de Neurologica La Fé University Hospital; Valencia
Locations (9):
- Aarhus University Hospital, Aarhus, Denmark
- Hospital Tenon Service de Neuro-urologie et d'Explorations Périnéales, Paris, France
- Italy (4):
  - Azienda Ospedaliero-Universitaria of Ferrara, Ferrara, Cona
  - AISM Liguria Rehabilitation Centre, Genoa, Liguria
  - AOU Careggi, Florence, Tuscany
  - Azienda Ospedaliero Universitaria Consorziale Policlinico con sede in Bari, Bari
- La Fé University Hospital, Valencia, Spain
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Switzerland
- University College London Hospital, London, United Kingdom